CLINICAL TRIAL: NCT05564026
Title: Pediatric Germ Cell Tumors: Outcomes, Genomics and Epigenetics
Brief Title: Molecular Epidemiology of Pediatric Germ Cell Tumors
Status: Recruiting | Type: Observational
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Other Study IDs: AEPI17N3
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Germ Cell Tumor; Germinoma; Teratoma; Embryonal Carcinoma; Yolk Sac Tumor; Choriocarcinoma; Mixed Germ Cell Tumor; Late Effects; Pediatric Germ Cell Tumor
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Germinoma; Teratoma; Carcinoma, Embryonal; Endodermal Sinus Tumor; Choriocarcinoma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Tumor Specimen Collection
  * Germline DNA Samples (saliva)
  * Blood Sample Collection (serum/plasma)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative: Children and adolescents with a germ cell tumor, previously enrolled on APEC14B1 or AEPI10N1 who allow access to medical records (including audiograms), grant permission to: evaluate of all of their DNA, place their genetic and health information in scientific databanks, and collect a blood sample at a routine clinic/home visit, as well as complete a questionnaire about your health and quality of life since treatment.
  Interventions: Other: Questionnaire Administration; Other: Tumor Specimen Collection; Other: Germline DNA Samples; Procedure: Blood Sample Collection

INTERVENTIONS:
Other: Questionnaire Administration — Questionnaire provide to participant's about their health and quality of life since treatment
Other: Tumor Specimen Collection — Tumor DNA requested from the Biopathology Center
Other: Germline DNA Samples — Germline DNA specimens requested from the Biopathology Center or newly collected saliva
Procedure: Blood Sample Collection — Collection and storing of serum/plasma

SUMMARY:
A Non-Therapeutic Study that aims to establish a cohort of GCT survivors to understand short term and long-term adverse effects of treatment and to conduct molecular analyses to improve risk stratification.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish a survivorship cohort for pediatric and adolescent GCT comprised of participants from AEPI10N1 and APEC14B1 to assess short term and long-term adverse events associated with GCT treatment.

II. Compare somatic variation by tumor histology to identify molecular signatures that improve prognostic risk stratification.

III. Identify methylation patterns that predict poor clinical outcomes, including disease relapse and death.

OUTLINE:

Medical records from pediatric and adolescent Germ Cell Tumor (GCT) participants from AEPI10N1 and APEC14B1 will be used to obtain treatment information and validate self-reported outcomes. Paired normal and tumor samples will be used to evaluate single nucleotide variants, indels, copy number variations, and DNA methylation patterns. Ototoxicity will be determined by central review of audiogram files obtained from the treating institutions and self-reported based on questionnaire data.

ELIGIBILITY:
Inclusion Criteria:

* Cases will be eligible for the study if they have a primary diagnosis of GCT including germinoma (ICCC code105 9060-9065), teratoma (9080-9084), embryonal carcinoma (9070-9072), yolk sac tumor (9071), choriocarcinoma (9100, 9103, 9104), and mixed GCT (9085, 9101, 9102, 9105) in all sites including the brain.
* The patient must be enrolled on APEC14B1 with consent to future contact or enrolled in AEPI10N1 with consent for future contact (N=827). Patients enrolled in AEPI10N1 were recruited from ACCRN07. All patients must be registered with COG by a North American member institution. Note: (history of) treatment on a COG therapeutic trial is not required.
* Patients must be diagnosed at < 20 years of age at the time of GCT diagnosis. Study participants will be followed over time in the survivorship study so there is no maximum age for participation.
* Participants must be able to complete study related documents in English or Spanish.
* All patients and/or their parents or legal guardians must provide informed consent. Assent will be obtained for participants between the ages of 8-17 years.
* All institutional, FDA, and NCI requirements for human studies must be met.

Exclusion Criteria:

* Participants from AEPI10N1 who did not consent to future contact. Patients who do not meet the eligibility criteria described above or cannot complete study materials in English or Spanish

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adolescent Germ Cell Tumor survivors recruited from recently completed Children's Oncology Group (COG) epidemiology study (AEPI10N1) and the COG Project:EveryChild Registry (APEC14B1).
Sampling Method: Non-Probability Sample
Enrollment: 1151 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Ototoxicity | Up to 5 years
  Ototoxicity as determined by central review of end of therapy audiograms will serve as the primary outcome variable for analyses. Current ototoxicity will be assessed using an app-based hearing assessment. For the app-based audiometry assessment, unilateral hearing loss will be defined as at least one pure tone threshold greater than 25 decibels across at any one of the frequencies from 2,000 Hz- 8,000 Hz to align with the SIOP Boston guidelines, while bilateral hearing loss will be defined as a pure tone threshold > 25 decibels in both ears at any one of the frequencies.
Somatic Mutations | Up to 5 years
  Compare somatic variation by tumor histology to identify molecular signatures that improve prognostic risk stratification. Somatic mutations will be identified by comparing tumor samples to normal samples. Risk stratification will be based on event free survival, defined as the time from diagnosis to relapse or death.
Methylation | Up to 5 years
  Compare the association between DNA methylation patterns and relapse or death. Mixed-effects regression models will be used to test for association between methylation beta values and poor outcomes. The outcome will be defined as a binary variable with a value of one if the patient experienced a relapse or death event and zero otherwise.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Poynter, PhD, Principal Investigator — Children's Oncology Group
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States